CLINICAL TRIAL: NCT06983938
Title: Randomized Trial Comparing Dual Perclose Vs Single Angioseal And Perclose in Patients Undergoing Transfemoral Transcatheter Aortic Valve Replacement
Brief Title: This Study Will Evaluate the Safety and Potential Complications of Dual ProGlide vs Single ProGlide and Angioseal for Common Femoral Arteriotomy Closure Following Transcatheter Aortic Valve Replacement
Acronym: TAVI-CLOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 024-458
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Transcatheter Aortic Valve Replacement; Closure Technique
Keywords: Transcatheter aortic valve replacement; Perclose Proglide; Angioseal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dual Perclose Proglide (Active Comparator): Upon completion of valve replacement, this cohort will be closed using dual Perclose Proglide devices.
  Interventions: Device: Double Perclose Proglide
- Single Perclose Proglide plus Angioseal (Active Comparator): Upon completion of valve replacement, this cohort will be closed using a single Perclose Proglide device and single Angioseal device.
  Interventions: Device: Single Perclose Proglide plus Angioseal

INTERVENTIONS:
Device: Double Perclose Proglide — Upon completion of valve replacement, closure will proceed using two Perclose Proglide devices.
  Arms: Dual Perclose Proglide
Device: Single Perclose Proglide plus Angioseal — Upon completion of valve replacement, closure will proceed using one Perclose Proglide device plus one Angioseal device.
  Arms: Single Perclose Proglide plus Angioseal

SUMMARY:
This prospective, randomized, parallel, single-center, open-label, non-inferiority study will evaluate the safety and potential complications of dual ProGlide vs single ProGlide and Angioseal for common femoral arteriotomy closure following Transcatheter Aortic Valve Replacement.

DETAILED DESCRIPTION:
This is a prospective, randomized, parallel, open-label, single-center, non-inferiority study.

Approximately 90 patients undergoing Transcatheter Aortic Valve Replacement with femoral access will be randomized in a 1:1 fashion to receive femoral access closure using either dual Perclose Proglide or single Perclose Proglide and Angioseal for closure.

The primary end point of this study is the composite endpoint of main access-related bleeding ≥Type 2 and main access related major vascular complication. Secondary end points include periprocedural complications (such as acute vessel closure, leg embolization and perforation), procedural characteristics (total duration, fluoroscopy time, contrast volume, length of hospital stay), and cost of hospitalization. A routine follow-up visit assessment will be performed at 30 days in the valve clinic and the assessment will include: any clinical change, re-interventions, and peripheral pulse evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Planned to undergo transcatheter aortic valve replacement via femoral access
* Able to provide written informed consent prior to study participation

Exclusion Criteria:

* Non-femoral access
* Previous repair or intervention of the common femoral artery
* Previous pseudoaneurysm of the common femoral artery
* Children below 18 years, prisoners, and patients who are unable to provide consent are excluded.
* In another research study that has not granted permission to dual-enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Main access-related bleeding and vascular complications | Periprocedural
  Primary endpoint collected will be composite endpoint of main access-related bleeding ≥Type 2 and main access related major vascular complication- VARC (Valve Academic Research Consortium) 3 Criteria.

SECONDARY OUTCOMES:
Periprocedural complications, procedural characteristics, hospitalization | Periprocedural through hospital discharge
  Secondary endpoints will be periprocedural complications, acute vessel closure, embolization, and vessel perforation, procedural characteristics (duration, fluoroscopy time, contrast volume), length of hospital stay, and cost of hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White The Heart Hospital - Plano, Plano, Texas, United States

REFERENCES:
- [Background] Kiramijyan S, Magalhaes MA, Ben-Dor I, Koifman E, Escarcega RO, Baker NC, Torguson R, Okubagzi P, Bernardo NL, Satler LF, Pichard AD, Waksman R. The adjunctive use of Angio-Seal in femoral vascular closure following percutaneous transcatheter aortic valve replacement. EuroIntervention. 2016 May 17;12(1):88-93. doi: 10.4244/EIJV12I1A16. PMID 27173868
- [Background] Ko TY, Kao HL, Liu YJ, Yeh CF, Huang CC, Chen YH, Hung CS, Chan CY, Lin LC, Chen YS, Lin MS. Intentional combination of ProGlide and Angio-Seal for femoral access haemostasis in transcatheter aortic valve replacement. Int J Cardiol. 2019 Oct 15;293:76-79. doi: 10.1016/j.ijcard.2019.05.055. Epub 2019 May 23. PMID 31155328
- [Background] Bazarbashi N, Ahuja K, Gad MM, Sammour YM, Kaur M, Karrthik A, Saad AM, Khubber S, Dhaliwal K, Mick SL, Navia JL, Puri R, Reed GW, Krishnaswamy A, Kapadia SR. The utilization of single versus double Perclose devices for transfemoral aortic valve replacement access site closure: Insights from Cleveland Clinic Aortic Valve Center. Catheter Cardiovasc Interv. 2020 Aug;96(2):442-447. doi: 10.1002/ccd.28585. Epub 2019 Nov 12. PMID 31713996